CLINICAL TRIAL: NCT04669444
Title: Investigation of Biomarkers, Genomics, Physiology in Critically Ill and ECMO Patients
Brief Title: Biomarkers, Genomics, Physiology in Critically Ill and ECMO Patients
Acronym: IGNITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Professor, Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 191464
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Distress Syndrome; Cardiac Failure; Extracorporeal Membrane Oxygenation Complication; Respiratory Failure; Renal Failure; Critical Illness; Pulmonary Disease
Keywords: ECMO; ARDS; Ventilator induced Lung Injury; Heart Failure; Pulmonary Failure; Biomarkers
MeSH Terms: conditions — Respiratory Distress Syndrome; Heart Failure; Respiratory Insufficiency; Renal Insufficiency; Critical Illness; Lung Diseases; Ventilator-Induced Lung Injury | interventions — Ventilators, Mechanical

STUDY DESIGN:
Intervention Model Description: Single group, intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Driving Pressure Protocol (Experimental): The patients ventilator driving pressure will be decreased (as tolerated by the patient) for 2 hours while on extracorporeal membrane oxygenation (ECMO) support.
  Interventions: Device: Ventilator

INTERVENTIONS:
Device: Ventilator — The patient starts at a ventilator driving pressure of 10-15 cm of H2O as per guidelines for patients on ECMO with ARDS. The driving pressure is then decreased as tolerated for two hours to evaluate the effects on pulmonary, cardiac, and inflammatory biomarkers.
  Other Names: Breathing Machine; Invasive mechanical ventilation

SUMMARY:
Patients in end-stage cardiac failure and/or respiratory failure may be started on a rescue therapy known as Extracorporeal Membrane Oxygenation (ECMO). One of the major clinical questions is how to manage the ventilator when patients are on ECMO therapy. Ventilator Induced Lung Injury (VILI) can result from aggressive ventilation of the lung during critical illness. VILI and lung injury such as Acute Respiratory Distress Syndrome (ARDS) can further increase the total body inflammation and stress, this is known as biotrauma. Biotrauma is one of the mechanisms that causes multi-organ failure in critically ill patients. One advantage of ECMO is the ability to greatly reduce the use of the ventilator and thus VILI by taking control of the patient's oxygenation and acid-base status. By minimizing VILI during ECMO we can reduce biotrauma and thus multi-organ failure. Since the optimal ventilator settings for ECMO patients are not known, we plan to study the impact of different ventilator settings during ECMO on patient's physiology and biomarkers of inflammation and injury.

ELIGIBILITY:
Inclusion Criteria

* Patient currently on ECMO (Veno-Venous or Venous-Arterial or Venous-Arterial-Venous)
* Patient that is a potential ECMO candidate.

Exclusion Criteria

* History of Lung or Cardiac Transplantation
* Patient is not committed to full support
* Treating clinician refusal, or unwillingness to commit to controlled ventilation for at least 4-6 hours (if patient is mechanically ventilated)
* Inability to get informed consent from the patient or surrogate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in plasma IL-6 level from baseline to low driving pressure ventilation | 2 hours
  IL-6 is a marker of systemic inflammation, previously used in studies of ECMO and ARDS.

SECONDARY OUTCOMES:
Change in plasma sRAGE from baseline to low driving pressure ventilation | 2 hours
  sRAGE is a marker of systemic inflammation and acute lung injury, previously used in studies of ECMO and ARDS.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Owens, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests for IPD will be considered by the investigators.